CLINICAL TRIAL: NCT01641757
Title: Effect of Non-Surgical Periodontal Therapy on Serum Albumin Levels of Patients on Maintenance Hemodialysis Therapy, A Randomized Control Trial
Brief Title: Effect of Non-Surgical Periodontal Therapy on Serum Albumin Levels of Patients on Maintenance Hemodialysis Therapy,
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of the Punjab (Other)
Responsible Party: Principal Investigator, Dr Arsalan Wahid, Principal Investigator, University of the Punjab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: arsalanmalik
Record Dates: First submitted 2012-07-10; First posted 2012-07-17 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: End Stage Renal Failure on Dialysis; Periodontitis
Keywords: hemodialysis; periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Dental Scaling; Root Planing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- periodontal treatment group (Experimental): non surgical periodontal therapy will be given to study subjects which will be selected by randomization from total study sample. at the end of study, serum albumin levels of both study and control groups will be compared.
  Interventions: Procedure: non-surgical periodontal therapy

INTERVENTIONS:
Procedure: non-surgical periodontal therapy — dental scaling and root planing of full mouth will be done
  Other Names: dental scaling and root planing

SUMMARY:
Periodontitis is a destructive chronic infection of the gums, ligaments, and bone, predominantly caused by Gram-negative bacteria. Individuals with periodontal disease are at increased risk of systemic diseases. Increased prevalence of periodontal disease has been reported in patients with chronic kidney disease, especially in dialysis patients. Chronic kidney disease (CKD) is the progressive loss of kidney function over time. When kidneys loose their 85-90 % function, dialysis is performed. Efficacy of dialysis is checked by serum albumin levels. Lower-than-normal levels of serum albumin may be a sign of kidney diseases. Hypoalbuminemia has been demonstrated to be a strong predictor of death in chronic renal failure. A proposed mechanism for the effect of periodontitis on the development of kidney disease is systemic inflammation. The deleterious effects of systemic inflammation on kidney function could occur during the period of active periodontal infection and accumulate during the life time of the individual. This randomized control trial is designed to observe the effect of non-surgical periodontal therapy on serum albumin levels of patients on maintenance hemodialysis therapy. Patients will undergo periodontal examination and their serum albumin levels will be checked. Then they will be randomly divided in two groups. One group will be given non surgical periodontal treatment and second group will be offered late treatment. After 6 weeks 1st group will be reevaluated by serum albumin level and periodontal examination to observe the effect of non-surgical periodontal therapy. Statistical analyses shall be performed using SPSS software. T tests and Chi-sq tests shall be used to test differences according to periodontal status for continuous and categorical variables, respectively. The level of significance is set at p<0.05.

DETAILED DESCRIPTION:
Periodontitis is a destructive chronic infection of the gums, ligaments, and bone, predominantly caused by Gram-negative bacteria residing in biofilm surrounding the teeth. Biofilm is an aggregate of microbes with a distinct architecture. This biofilm contains clusters of bacterial species that are found commonly below the gingiva and are associated reproducibly with periodontal disease. These bacteria involved in periodontitis causes destruction of tissues which leads to formation of a periodontal pocket. This space becomes a site for further bacterial colonization and possible entry route of bacteria in blood stream.

It is evident from the data that periodontal health of the Pakistani nation is very poor with only 28% of the 12 year old having healthy gums and more than 93% of the 65 year old have some gum or periodontal disease . These results indicate that periodontal disease including inflammation of gums and calculus is endemic in Pakistan . Like caries, the level of gingival and periodontal disease is higher in the rural population of the Pakistan.

There is an increasing evidence that individuals with periodontal disease are at increased risk of cardiovascular disease, preterm delivery of low birth weight infants, pulmonary diseases, diabetes, osteoporosis, rheumatoid arthritis, alzheimer's disease & kidney diseases. The factors predisposing to periodontal disease and accelerating its progression are clearly evident in chronic renal failure. They encompass hyposalivation and xerostomia, impaired immunity and wound healing, alveolar bone destruction due to renal osteodystrophy, bleeding diathesis, diabetes mellitus, malnutrition and a state of general disability impairing oral hygiene. There is evidence for increased prevalence of periodontal disease in patients with renal disease, especially in dialysis patients.

Chronic kidney disease (CKD) is the progressive loss of kidney function over time. Normal renal functions are normally evaluated by glomerular filtration rate (GFR). Normal results range from 90 - 120 mL/min/1.73 m2.

The loss of kidney function usually takes months or years to occur. The final stage of chronic kidney disease is called end-stage renal disease (ESRD) after which kidneys no longer function and the patient needs dialysis or a kidney transplant .

Chronic kidney disease changes the serum levels of Albumin, Potassium, Calcium, Phosphorus, Sodium, Cholesterol and electrolytes. Among all these, albumin is of prime importance because it plays an important role in keeping the fluid from the blood from leaking out into the tissues. The normal range is 3.4 - 5.4 grams per deciliter (g/dL).

Lower-than-normal levels of serum albumin may be a sign of kidney diseases or liver disease (for example, hepatitis, cirrhosis). Decreased albumin may occur when body does not get or absorb enough nutrients, such as after Crohn's disease, Low-protein diets, Sprue, Whipple's disease . Other conditions under which the albumin levels are need to be measured are widespread burns and Wilson,s disease.

Hypoalbuminemia has been demonstrated to be a strong predictor of death in chronic renal failure . Some studies have however suggested that hypoalbuminemia may be more indicative of underlying inflammation, rather than nutritional status, especially in patients with kidney disease. In a study it was observed that on dialysis initiation in the US pediatric population, hypoalbuminemic patients were at higher risk of dying as compared to patients in whom dialysis was initiated with normal albumin levels . It was also assessed that hypoalbuminemia, is highly prevalent in kidney failure and is associated with an increased mortality risk in this population. Serum albumin level may reflect both the nutritional status and chronic inflammation.

A proposed mechanism for the effect of periodontitis on the development of kidney disease is systemic inflammation . Periodontal pathogens have been shown to have the ability to adhere to, invade, and proliferate in coronary endothelial cells leading to atheroma formation and impaired vasculature relaxation. Cardiovascular diseases and CKD share many risk factors, so it is it can be assumed that periodontal disease exerts similar effects within the vasculature of the kidney. Both periodontitis and kidney diseases are associated with inflammatory markers such as C-reactive protein and chronic low level inflammation associated with periodontitis may lead to endothelial dysfunction which plays a role in the pathogenesis of kidney disease in edentulous patients. The deleterious effects of systemic inflammation on kidney function could occur during the period of active periodontal infection and accumulate during the life time of the individual. Inflammation is an important predictor of low serum albumin levels among dialysis patients, independent of nutritional status. Low albumin is often indicative of malnutrition, but chronic inflammation appears to be the culprit in half of the patients with low levels of albumin. This may explain why nutritional therapy does not increase serum albumin levels in some patients suggesting chronic inflammation. High CRP levels correlates with increased mortality, regardless of nutritional status suggesting an independent role for chronic inflammation in causing hypoalbuminemia .

Abhijit V. Kshirsagar et al. observed an association of severe periodontal disease and hypoalbuminemia in a group of patients who were receiving long-term outpatient hemodialysis. In study subjects, patients with periodontal disease were more than three times more likely to have low serum albumin than patients without periodontal disease. Increased levels of plaque have been reported for hemodialysis (HD) populations from several countries including Brazil. It has to be noted, however, that HD patients are also repeatedly exposed to systemic anticoagulation with high-dose heparin during blood purification procedures. This predisposes them further to gingival bleeding and, in consequence, facilitates bacterial colonization and growth, and may propagate periodontal disease. Recently, an impressive 3-fold decrease in C-reactive protein and a rise in hemoglobin (Hb) levels in HD patients were reported to occur already after 4-6 weeks following traditional periodontal therapy . Thus, the issue of poor oral health status in CKD patients apparently deserves a higher awareness of the problem, and increased attention, and indicates the need for a closer collaboration between primary care physicians, nephrologists and dentists.

There is evidence supporting the contribution of periodontitis to systemic inflammation. Several possible mechanisms have been suggested, including the locally produced inflammatory mediators and bacterial by-products that invade the blood stream, interact with host cells and trigger inflammatory response.

A study from Turkey of End Stage Renal disease (ESRD) patients on HD therapy found increased periodontitis as measured by the Community Periodontal Index of Treatment Needs (CPITN). In a study of renal patients receiving HD, Chaung et al, 2005 in Taiwan, reported increased rates of periodontitis when compared with national data on periodontal disease for the Taiwanese population. Studies focusing on the periodontal health of End Stage Renal disease (ESRD) patients on HD maintenance therapy have reported the presence of poor oral hygiene and attendant gingival inflammation.

Bots CP, Poortermann JHG, Brand HS et al (2006) in a study from Netherlands of ESRD patients, some of whom were receiving HD, did not find an increased loss of attachment when compared with some healthy case-matched controls. Periodontal status of End stage Renal Disease (ESRD) patients receiving HD showed no increase in periodontal indices when compared with case-matched controls. The authors did note that the HD group had greater numbers of periodontopathic bacterial species than the control group.

The results of studies conducted so far to establish association between severe periodontitis and hypoalbuminemia are variable and are not conclusive. Only one clinical trial has been conducted regarding that, therefore aim of the study is to observe the effect of non surgical periodontal therapy on changes of albumin levels in maintenance dialysis patients.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic Kidney Disease patients, who are receiving hemodialysis therapy for >3 months. of all ages and both gender and are able to give informed consent.
2. Have at least 14 teeth (excluding third molars) in oral cavity shall be included in study.

Exclusion Criteria:

1. Patients have had periodontal therapy <1 year.
2. Diabetes Mellitus
3. Liver disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2012-05; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
serum albumin levels | 6 months
  serum albumin levels are considered to be strong predictor of death in dialysis patients. in this trial we want to see the effect of non surgical periodontal therapy on serum albumin levels of patients on maintenance dialysis therapy

CONTACTS AND LOCATIONS:
Overall Officials: Ayyaz A Khan, PhD, Study Director — Shaikh Zayed Medical CompleX lahore
Locations (1):
- Shaikh Zayed Medical Complex, Lahore, Punjab Province, Pakistan

REFERENCES:
- [Background] Bots CP, Poorterman JH, Brand HS, Kalsbeek H, van Amerongen BM, Veerman EC, Nieuw Amerongen AV. The oral health status of dentate patients with chronic renal failure undergoing dialysis therapy. Oral Dis. 2006 Mar;12(2):176-80. doi: 10.1111/j.1601-0825.2005.01183.x. PMID 16476040